CLINICAL TRIAL: NCT01176786
Title: The Effect of Reusable Versus Disposable Draping on Implant Based Breast Reconstruction Infection Rates: a Prospective Randomized Study
Brief Title: Reusable Versus Disposable Draping System in Breast Reconstruction Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 10667
Record Dates: First submitted 2010-08-05; First posted 2010-08-06 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-06

CONDITIONS: Mastectomy; Infections; Breast Reconstruction
Keywords: infection; tissue expander; breast implant; breast reconstruction; Infections rates
MeSH Terms: conditions — Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Culture Swabs, Rodac Plate Cultures — Culture swab is taken when breast tissue expander is removed and when breast implant is placed in breast pocket. Rodac Plate cultures are taken after the surgical procedure of the surgeons dominant palm, forearm of gown and subject's drape closest to the breast.

SUMMARY:
This study will look at the rate of infections developed by subjects comparing the use of disposable draping systems versus reusable draping systems in the operating room.

DETAILED DESCRIPTION:
Subjects enrolled in the study will be randomized into two groups. One group will have the reusable draping system during surgery which the investigators currently use and the second group will have the disposable draping system. Subjects will be blinded to the type of draping system used. Subjects are under anesthesia at the time the surgical drapes are placed. After the subject has signed the informed consent, they will be assigned a study number for that surgery. The study number will correlate to an envelope which will contain information on the type of draping system to be used. Subjects enrolled, may be randomized more than once. Subjects will typically have a minimum of two surgeries, the placement of the tissue expanders and then the removal of the expanders and placement of the breast implants. Subjects will not be required to sign another consent form but will be randomized prior to each surgery. Surgeons who have subjects in the disposable draping system will use a disposable draping kit that includes gowns for the surgeons and also towels. For subjects who are having a mastectomy and then the placement of tissue expanders, after the mastectomy has been performed, the plastic surgeons will use all new draping, towels and gowns to perform tissue expander placement. A swab will be taken on the wound site to determine if there are any CFUs (colony forming units) present. The swab will then be placed in a tube containing 1ml of TSB (triptic soy broth). The tube will then be sonicated , and then vortexed for 15 seconds. A 0.1ml aliquot of the solution will be placed in a blood agar plate and incubated for 48 hours to determine the CFU count. The remainder of the solution will be frozen. In the event an infection occurs, molecular matching will be done on the culture to determine if it is from the same exact culture. Rodac plates will be used to test for the presence of bacterial cultures on the surgeon's gown (Forearm [volar surface]) and glove (palm of surgeon's dominate hand) and also the subject's surgical drape (Area over sternum). These will be incubated for 48 hours to determine the CFU count. This process will be repeated at the second surgery.

ELIGIBILITY:
Inclusion Criteria:

Females ages 18 years of age and older who are having a mastectomy with tissue expander placement and for breast implants for reconstruction, which would include immediate or delayed reconstruction.

Exclusion Criteria:

Male subjects are excluded from this study, while some males do have breast cancer, this is a rare occurrence and they do not undergo reconstruction surgery with expanders and breast implants. Females under the age of 18 are excluded as well as females who undergo a mastectomy but do not have any reconstruction surgery. Females who otherwise meet the criteria but have an active infection, currently on antibiotics to treat an infection, urinary tract infections, soft tissue infections or pneumonia are also excluded until they are approved for surgery by the physician.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2009-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Infection rates of reusable versus disposable draping system in the operating room | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Lisa David, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Baptist Medical Center Plastic & Reconstructive Surgery Department, Winston-Salem, North Carolina, United States